CLINICAL TRIAL: NCT05200364
Title: A Phase 1 Open-Label, Safety, Pharmacokinetic and Preliminary Efficacy Study of STRO-002, an Anti-Folate Receptor Alpha Antibody Drug Conjugate, in Combination With Bevacizumab in Patients With Advanced Epithelial Ovarian Cancer (Including Fallopian Tube or Primary Peritoneal Cancers)
Brief Title: A Study of STRO-002, an Anti-Folate Receptor Alpha Antibody Drug Conjugate, in Combination With Bevacizumab in Epithelial Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated Early
Sponsor: Sutro Biopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STRO-002-GM2
Record Dates: First submitted 2021-12-19; First posted 2022-01-20 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer; Ovarian Carcinoma; Ovary Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: The study is designed as a 3+3 dose escalation/de-escalation of STRO-002 given in combination with the labeled dose of bevacizumab. The patient population is relapsed ovarian cancer and the study treatment is the combination of STRO-002 plus bevacizumab. This study will be conducted in 2 parts, dose escalation and dose expansion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental :STRO-002 treatment in combination with Bevacizumab (Experimental): Dose Escalation: STRO-002 at increasing dose levels plus bevacizumab at 15 mg/kg
  Dose Expansion: STRO-002 at RP2D plus bevacizumab at 15 mg/kg
  Interventions: Drug: STRO-002; Drug: Bevacizumab

INTERVENTIONS:
Drug: STRO-002 — intravenous antibody drug conjugate
Drug: Bevacizumab — anti-VEGF agent
  Other Names: Avastin

SUMMARY:
Phase 1 trial to study the safety, pharmacokinetic and Preliminary Efficacy of STRO-002 in combination with Bevacizumab.

DETAILED DESCRIPTION:
This study is a Phase 1, open-label, multicenter, dose escalation study to assess preliminary efficacy for STRO-002 combined with bevacizumab in patients with advanced ovarian cancer that is refractory or has relapsed after standard available therapy. Fallopian tube and primary peritoneal cancers are treated in the same manner as epithelial ovarian cancers and are thus included in this study.

The dosing regimen will include bevacizumab administered at the labeled dose of 15 mg/kg IV q 3 weeks given together with STRO-002 at increasing dose levels administered IV q 3 weeks. The RP2D of STRO-002 given with bevacizumab 15 mg/kg q 3 weeks will be determined by dose escalation.

Dose expansion will enroll approximately 40 subjects with advanced relapsed ovarian cancer treated with STRO-002 plus bevacizumab at the RP2D determined in dose escalation. Subjects in the dose expansion portion of the study will be required at screening to submit both archival tumor tissue (if available and available tissue has adequate tumor) and tumor tissue from a biopsy done during screening to the central laboratory for analysis of FOLRα expression, both prior to enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. ECOG 0-1
3. Life expectancy > 3 months
4. High Grade serous epithelial ovarian cancer (EOC), fallopian tube or primary peritoneal cancer with pathology report documentation of tumor type.
5. At least one measurable target lesion per RECIST v1.1.
6. Tumor tissue for FolRα expression testing prior to enrollment.

   1. For dose escalation: tissue may be from either archival tumor tissue or from a biopsy performed during screening.
   2. For dose expansion part of the study, tissue from both archival tumor tissue and a biopsy performed during screening is required.
7. Adequate bone marrow function defined as:

   1. Absolute neutrophil count (ANC) ≥1500/μL
   2. Hemoglobin ≥ 9g/dL
   3. Platelet count ≥ 100 x 10^3/μL
8. Adequate liver function defined as:

   1. ALT and AST < 2.5 x ULN
   2. ALP < 2.5 x ULN
   3. Bilirubin < 1.5 x ULN
9. Adequate renal function defined as serum creatinine ≤ 1.5 x ULN or creatinine clearance (CrCl) > 40 mL/min.

   Subjects enrolling into Dose Escalation must also meet the following inclusion criteria:
10. Relapsed and/or PD on last treatment regimen and one of the following:

    1. Primary Platinum refractory and received no more than 1 prior regimen
    2. Primary platinum resistant and received no more than 4 prior regimens
    3. Platinum sensitive and all of the following:

       * received at least 2 platinum-based therapies or received 1 platinum and 1 non-platinum based therapy (if unable to receive a second platinum regimen due to toxicity) or received at least 1 platinum-based therapy (if the regimen contained a PARP inhibitor given as maintenance treatment)
       * received no more than 1 additional regimen after becoming platinum resistant
       * received no more than 4 prior regimens

    Subjects enrolling into Part 2, Dose Expansion must also meet the following inclusion criteria:
11. Relapsed and/or PD on last treatment regimen and one of the following:

    1. Platinum resistant and received no more than 4 prior regimens
    2. Platinum sensitive and

       * received at least 2 platinum-based therapies or received 1 platinum and 1 non-platinum based therapy (if unable to receive a second platinum regimen due to toxicity) or received at least 1 platinum-based therapy (if the regimen contained a PARP inhibitor given as maintenance treatment)
       * received no more than 1 additional regimen after becoming platinum resistant
       * received no more than 4 prior regimens

Exclusion Criteria:

1. Low grade ovarian carcinoma (Grade 1).
2. Clear cell, mucinous, endometrioid, sarcomatous, and mixed histology ovarian carcinomas, endometrial leiomyosarcoma, and endometrial stromal sarcomas.
3. Prior treatment with an ADC with a tubulin inhibitor warhead.
4. Prior treatment with other FolRα targeting agents unless approved by a Sutro medical monitor or designee.
5. Subjects who are primary platinum-refractory during frontline treatment are excluded from the Expansion Cohort (Allowed in Dose Escalation if no more than 1 prior regimen).
6. Greater than 4 prior lines of treatment (> 1 prior if primary platinum refractory).
7. Any prior toxicity that required permanent discontinuation of bevacizumab or other contraindication to receive bevacizumab per institutional guidelines.
8. Previous solid organ transplantation.
9. Current signs/symptoms of bowel obstruction and/or signs/symptoms of or bowel obstruction within 3 months of initiation of study treatment.
10. Grade ≥2 toxicity from prior anticancer therapy with the exception of Grade 2 alopecia or Grade 2 neuropathy.
11. Uncontrolled hypertension
12. Sensory or motor neuropathy Grade > 1 at screening prior to initiation of study treatment.
13. Potentially fatal concurrent or recent malignancy. Subjects with past or current malignancy need to be discussed with the sponsor to determine eligibility.
14. Chronic or ongoing active infection requiring systemic treatment.
15. Ongoing immunosuppressive therapy, including systemic corticosteroids. Note: Physiologic replacement and use of topical or inhaled corticosteroids are allowed. Dexamethasone may be used to treat chemotherapy induced nausea per institutional guidelines.
16. Clinically significant cardiac disease.
17. History or clinical signs of meningeal or active central nervous system involvement.
18. Known severe COPD or asthma
19. Active pneumonitis within 6 months of initiating study treatment.
20. History of stroke or history of significant cerebrovascular disease (i.e., transient ischemic attack) within 6 months of initiation of study treatment.
21. History of pulmonary embolism or any Grade 3 thromboembolic event within 6 months of initiation of study treatment.
22. Known human immunodeficiency virus seropositivity.
23. Active hepatitis B or hepatitis C and positive serology (unless due to vaccination or passive immunization due to immunoglobulin therapy) with the following exceptions:

    1. Subject has had HCV but received antiviral treatment and shows no detectible HCV viral DNA for 6 months prior to screening
    2. Subject has had HBV but is HBV surface antigen (HBsAg) and viral DNA negative at screening
    3. Subject has had HBV but received antiviral treatment and have undetectable viral DNA for 6 months prior to screening
24. Concurrent participation in another therapeutic treatment trial
25. Significant concurrent, uncontrolled medical condition including, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral or psychiatric disease
26. Females who are pregnant or breastfeeding, and all women of childbearing potential unwilling to use adequate barrier contraception while on treatment and for 16 weeks after last dose of STRO-002/bevacizumab and 6 months after the last dose of bevacizumab.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients are required to have ovarian, fallopian, or primary peritoneal cancer.
Enrollment: 58 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Part 1 - Safety and tolerability of STRO-002/bevacizumab as a combination therapy | From baseline through end of study (approximately 24 months)
  Incidence and severity of adverse events (AEs) and clinical laboratory abnormalities observed across STRO-002/bevacizumab dose levels. Incidence of dose-limiting toxicities (DLTs) through Day 1-21 following administration of each initial STRO-002/bevacizumab dose.
Part 1 - Determine the recommended phase 2 dose (RP2D) of STRO-002/bevacizumab | From baseline through end of study (approximately 24 months)
  Frequency of DLTs across STRO-002 dose levels

SECONDARY OUTCOMES:
Part 1 - Characterize the pharmacokinetics (PK) of STRO-002 by measuring the maximum plasma concentration (Cmax). | From baseline through end of study (approximately 24 months)
  Measurement of maximum plasma concentration (Cmax) after the administration of STRO-002
Part 1 - Characterize the PK of STRO-002 by measuring the area under the plasma concentration versus time curve (AUC) | From baseline through end of study (approximately 24 months)
  Measurement of AUC
Part 1 - Assess the formation of anti-drug antibodies (ADAs) to STRO-002 when administered with bevacizumab. | From baseline through end of study (approximately 24 months)
  Circulating ADAs formed to STRO-002

CONTACTS AND LOCATIONS:
Overall Officials: Arturo Molina, MD, Study Chair — Sutro Biopharma
Locations (6):
- United States (6):
  - University of South Florida,, Tampa, Florida
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Li X, Zhou S, Abrahams CL, Krimm S, Smith J, Bajjuri K, Stephenson HT, Henningsen R, Hanson J, Heibeck TH, Calarese D, Tran C, Yin G, Stafford RL, Yam AY, Kline T, De Almeida VI, Sato AK, Lupher M, Bedard K, Hallam TJ. Discovery of STRO-002, a Novel Homogeneous ADC Targeting Folate Receptor Alpha, for the Treatment of Ovarian and Endometrial Cancers. Mol Cancer Ther. 2023 Feb 1;22(2):155-167. doi: 10.1158/1535-7163.MCT-22-0322. PMID 36459691